CLINICAL TRIAL: NCT01898286
Title: Open-Label Study to Evaluate Long Term Safety and Treatment Effect of DiaPep277® in Subjects Who Have Completed Study 1001 (NCT01103284)
Brief Title: Open-Label Extension Study to Evaluate Long Term Safety and Treatment Effect of DiaPep277®
Acronym: DIA-AID 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A corporate decision to suspend development of DiaPep277®
Sponsor: Andromeda Biotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1010; 2013-002775-17 (EudraCT Number)
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes
Keywords: C peptide; beta cell function; immune modulation of type 1 diabetes; immune intervention in type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DiaPep277® (Experimental): Administration of DiaPep277® to patients previously enrolled in the Phase 3 Study 1001 (NCT01103284)
  Interventions: Drug: DiaPep277®

INTERVENTIONS:
Drug: DiaPep277® — 1 mg of DiaPep277® subcutaneously in the upper arm at 0, 3, 6, 9, 12, 15, 18, and 21 months, for a total of 8 administrations

SUMMARY:
This is an extension study to evaluate the safety and tolerability of long-term treatment with DiaPep277® and to determine the long-term treatment effect of DiaPep277® on parameters of metabolic control and on preservation of beta-cell function in subjects who have long exposure to DiaPep277®.

DETAILED DESCRIPTION:
Treatment with DiaPep277® is expected to be long-term; stopping treatment may result in the eventual loss of the preserved beta-cell function. Indeed, extension of phase 2 studies has shown that patients who were initially treated with DiaPep277® and maintained their initial beta-cell function, required continuation of treatment, losing beta-cell function if switched to Placebo. These extension studies were too small for the outcome to be statistically significant, but they suggested that continuation of treatment is needed for long-term maintenance of efficacy.

Therefore, in this extension study, patients who complete the 1001 phase 3 study (NCT01103284) and maintain clinically significant beta-cell function are offered a 2-year continuation of active treatment, since they are likely to benefit from use of the medication. The participation in the extension study will be offered to all eligible subjects who complete the 1001 study, regardless of the treatment arm allocation in the initial study.

By achieving long-term preservation of beta-cell function, patients are expected to maintain good management of the disease, manifesting as better glycemic control and fewer hypoglycemic events.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 1 diabetes who participated in the 1001 study
* residual beta-cell function demonstrated by stimulated C-peptide ≥ 0.20 nmol/L.

Exclusion Criteria:

* The subject has any significant ongoing diseases or conditions that is likely to affect the subject's response to treatment
* The subject has a history of any kind of malignant tumor.
* The subject has clinical evidence of any diabetes-related complication
* Subject has history of endogenous allergic reactivity:
* The subject has a known immune deficiency

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Raz, MD, Principal Investigator — Hadassah Medical Center, Jerusalem
Locations (3):
- United States (3):
  - Atlanta Diabetes associates, Atlanta, Georgia
  - Henry Ford Medical Centers - New Center One, Detroit, Michigan
  - Mountain Diabetes and Endocrine Center, Asheville, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients diagnosed with Type 1 diabetes mellitus up to six months before randomization to Study 1001 (NCT01103284), from medical sites in the EU, US, Russia, and Israel
Groups:
- Patients Treated With DiaPep (Originally Enrolled in Study1001: All patients enrolled in the 1010 study (NCT01898286), whether previously treated with DiaPep277 or placebo in the 1001 study (NCT01103284).
Period: Overall Study
Arm/Group | Patients Treated With DiaPep (Originally Enrolled in Study1001
Started | 38
Completed | 35 (For this study "completed" is defined as completing the Early Termination visit)
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients Treated With DiaPep (Originally Enrolled in Study1001
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.16 (7.343)
Age, Customized [Median (Full Range); unit: years] | 32.00 [23.0 to 47.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 33
  Hispanic | 1
  Black | 3
  Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemic Events
Description: The number of hypoglycemic events recorded by each patient over the course of the study.
Time Frame: At Early Termination Visit, Up to 25 Months
Population: Patients with hypoglycemic event data at the time of their early termination visit. This population is smaller than the population numbers in the patient flow categories because not all patients were willing to provide information on hypoglycemic events at early termination.
Measure: Mean (Standard Deviation); unit: hypoglycemic events
Arm/Group | Patients Treated With DiaPep (Originally Enrolled in Study1001
Number analyzed (Participants) | 16
hypoglycemic events | 3.3 (3.30)

2. Secondary Outcome: Change From Baseline in Glucagon-stimulated C-peptide AUC at Early Termination Visit
Description: Beta-cell function, measured as change in stimulated C-peptide secretion measured 0, 2, 6, 10 and 20 minutes post administration [area under the curve (AUC), 0-20 minutes] at Baseline and the early termination visit (up to 25 months), during a glucagon stimulation test (GST). Change was calculated for each patient by subtracting the baseline AUC value (defined as the last non-missing assessment prior to first dose in the 1010 study but after the end of study 1001) from the early termination visit AUC.
Time Frame: Baseline and Early Termination Visit, Up to 25 Months
Population: Only 9 patients had sufficient data for this analysis, as many patients declined to undergo the GST at the termination visit.
Measure: Mean (Standard Deviation); unit: nmol*minute/L
Arm/Group | Patients Treated With DiaPep (Originally Enrolled in Study1001
Number analyzed (Participants) | 9
nmol*minute/L | 0.2 (2.334)

3. Other Pre Specified Outcome: Change From Baseline in Daily Insulin Dose, Per kg Body Weight, at Early Termination Visit
Time Frame: Baseline and Early Termination Visit, up to 25 months
Population: All patients with daily insulin dose data at baseline and their early termination visit. Only 11 patients could be included in this analysis, as not all patients provided insulin dose data at their early termination visit.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Patients Treated With DiaPep (Originally Enrolled in Study1001
Number analyzed (Participants) | 11
IU/kg | 0.025 (0.0270)

4. Other Pre Specified Outcome: Glycemic Control (Change From Baseline in % HbA1c)
Time Frame: Baseline and Early Termination Visit, Up to 25 Months
Population: All patients with % HbA1c data at baseline and their early termination visit. Only 5 patients were available for this analysis, as not all patients agreed to complete HbA1c testing at the early termination visit.
Measure: Mean (Standard Deviation); unit: % HbA1c
Arm/Group | Patients Treated With DiaPep (Originally Enrolled in Study1001
Number analyzed (Participants) | 5
% HbA1c | 0.46 (0.907)

ADVERSE EVENTS:
Time Frame: AE data were collected from the time of subject enrollment through each subject's early termination visit
Arm/Group | Patients Treated With DiaPep (Originally Enrolled in Study1001
Serious Adverse Events (participants affected / at risk) | 1/38
Other Adverse Events (participants affected / at risk) | 9/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With DiaPep (Originally Enrolled in Study1001 (N=38)
Anaphylaxic shock for glucagon (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With DiaPep (Originally Enrolled in Study1001 (N=38)
Nasopharyngitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Electrocardiogram QT prolonged (Investigations) | 2
Blood cholesterol increased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Urine albumin/creatinine ratio increased (Investigations) | 1
Injection site erythema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Anxiety (Psychiatric disorders) | 1
Social phobia (Psychiatric disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Syncope (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
The objectives of this study were to evaluate the safety and tolerability of long term treatment with DiaPep277. The study was terminated by the Sponsor on 08Sep14; hence many of the protocol-specified objectives could not be adequately assessed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall submit any paper or presentation to the Sponsor for review and comments at least 60 days prior to submitting the same to a third party. Upon receiving any request from the Sponsor to delete any Confidential Information or request to delay in publication up to 90 days to allow the filing of any Sponsor application, the Investigator shall take the request action. Investigator shall not be restricted after 18 months from completion of their site's performance in the study.